CLINICAL TRIAL: NCT00969059
Title: A Randomised, Double Blind Study to Evaluate the Safety and Efficacy of the p38 Kinase Inhibitor, GW856553, in Subjects With Neuropathic Pain From Peripheral Nerve Injury
Brief Title: Study in Neuropathic Pain Patients With Peripheral Nerve Injury
Acronym: PNI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112967
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Pain, Neuropathic
Keywords: peripheral nerve injury; p38 kinase inhibitor; neuropathic pain
MeSH Terms: conditions — Neuralgia; Peripheral Nerve Injuries | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLACEBO (Placebo Comparator): Eligible participant with at least moderate intensity of pain (an average daily pain score of ≥ 4 on the 11 point PI-NRS at baseline) will receive placebo for 28 days.
  Interventions: Drug: PLACEBO
- Active (Experimental): Eligible participant with at least moderate intensity of pain (an average daily pain score of ≥ 4 on the 11 point PI-NRS at baseline) will receive 7.5 mg twice daily (bid) GW856553 for 28 days.
  Interventions: Drug: GW856553

INTERVENTIONS:
Drug: GW856553 — GW856553 is a film coated white tablet, 9mm round, biconvex, plain faced. It will be administered 7.5mg bid, orally with food at breakfast and dinner.
  Arms: Active
Drug: PLACEBO — Matching Placebo is a film coated white tablet, 9mm round, biconvex, plain faced. It will be administered orally with food at breakfast and dinner.
  Arms: PLACEBO

SUMMARY:
This study will be a double-blind, placebo-controlled, parallel group study. After enrolment and initial assessments, subjects will receive oral GW856553 7.5 milligram (mg) twice daily (BID) or matching placebo for 28 days in a 1:1 ratio. Sufficient numbers of subjects will be recruited to obtain 142 evaluable subjects. This is a double-blind, randomized, placebo-controlled, parallel group study. Subjects will undertake a screening period which may last up to approximately 3 weeks, followed by a baseline period of 1 week, a randomized treatment period of 4 weeks and a follow-up period of approximately 2 weeks. This is a multi-centre, double-blind, randomized, placebo-controlled study in subjects who have at least moderate intensity of neuropathic pain resulting from peripheral nerve injury due to trauma or surgery. It will investigate the efficacy, safety and tolerability of GW856553 over 28 days of treatment. Approximately 158 subjects will be randomized to ensure 142 evaluable subjects. Randomization ratio will be 1:1 for placebo or GW856553 respectively. The dose of GW856553 will be 7.5 mg BID.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 - 80 years inclusive, at the time of signing the informed consent.
* Female of non-child bearing potential or child bearing potential who agrees to use appropriate contraception methods.
* A diagnosis of peripheral neuropathic pain
* Focal neuropathic pain related to nerve injury caused by trauma or surgery not associated with an acute medical condition or injury by avulsion (examples include but are not limited to neuropathic pain secondary to surgical procedures such as thoracotomy, mastectomy, inguinal herniorrhaphy and radical neck dissection, traumatic mononeuropathies and brachial plexus or lumbosacral injuries due to bullet wounds, lacerations, road traffic accidents etc).
* Location of pain consistent with the area innervated by the affected nerve(s), with or without other sensory symptoms in the affected area.
* Duration of pain should be at least 12 weeks since the initial insult.
* Subjects on medications for neuropathic pain (including tricyclic antidepressants, anticonvulsants, opioids, tramadol, bupropion, venlafaxine, mexiletine, muscle relaxants, N-methyl-D-aspartate (NMDA) antagonists) but excluding but excluding non-steroidal anti-inflammatory drugs (NSAIDs), cycloxygenase-2 inhibitors (COX-2) , topical lidocaine, topical capsaicin, nerve blocks and steroid injections may only be included in the study if they have been on stable doses of such medications for at least 4 weeks prior to baseline period (Day -7).
* Participants who have been on NSAIDs, COX-2 inhibitors and topical lidocaine may only be included in the study if they have stopped these medications for at least 5 half-lives prior to the baseline period (Day -7). In the case of topical capsaicin, subjects should have stopped this for at least 8 weeks prior to the baseline period.
* Participants who have received nerve blocks or steroid injections for neuropathic pain may be included if their most recent treatment was at least 4 weeks prior to the baseline period (Day -7).
* Subjects' baseline average daily pain score on the PI-NRS, calculated as the average of their daily PI-NRS scores over the 7 days prior to Day 1, is greater than or equal to 4 on the PI-NRS, after wash-out of prohibited medications. Subjects will need to have recorded their daily PI-NRS for a minimum of 4 days during the 7 days prior to Day 1. Subjects will not be told prior to the completion of the baseline period that the entry requirement of the average PI-NRS is at least 4, in order not to bias their pain intensity score during the baseline period.
* Male subjects must agree to use appropriate contraception methods.
* Body weight >=50 kg for men and >=45 kg for women.
* Participants has provided full written informed consent prior to the performance of any protocol-specified procedure, which includes compliance with the requirements and restrictions.
* Single QT duration corrected for heart rate by Bazett's formula (QTcB) or QT duration corrected for heart rate by Fridericia's formula (QTcF) < 450 msec; or QTc < 480 milliseconds (msec) in subjects with Bundle Branch Block. If the first QTc exceeds the above limits, repeat the ECG twice at least 5 min apart and take the mean of the three QTc values to determine that the mean QTc satisfies the above limits.
* A subject with a clinical abnormality or other laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

Exclusion Criteria:

* Subjects with other causes for their neuropathic pain [e.g. trigeminal neuralgia, painful diabetic neuropathy, mononeuritis multiplex, central post-stroke pain, failed back surgery, phantom limb pain, peripheral neuropathy due to alcoholism, malignancy, human immunodeficiency virus (HIV), syphilis, drug abuse, cobalamin (vitamin B12) deficiency, hypothyroidism, liver disease, toxic exposure], substantial somatic pain component or more than one cause or potential cause for pain symptoms or nerve entrapment or chronic neck or back pain of more than mild degree or any concurrent rheumatic disease such as but not limited to fibromyalgia or rheumatoid arthritis.
* Subjects with intractable pain of unknown origin or active infection/inflammation in the area of nerve injury.
* Subjects who have had extensive soft tissue injury associated with extensive surgery in the treatment of their nerve injury. Any question regarding the definition of extensive surgery should be discussed with the GSK medical monitor.
* A positive pre-study drug/alcohol screen. However, a positive drug screen will not automatically exclude a subject if there is a medical explanation for the positive result other than drug abuse e.g. a subject who is taking opioids for their neuropathic pain.
* A positive test for HIV antibody.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* History of any liver disease within the last 6 months.
* History of excessive regular alcohol consumption within 6 months of the study.
* History or presence of significant cardiovascular, gastro-intestinal, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs which, in the opinion of the Investigator may interfere with the study procedures or compromise subject safety.
* History or presence of any clinically significant abnormality in vital signs / ECG / laboratory tests, or have any medical or psychiatric condition, which, in the opinion of the Investigator, may interfere with the study procedures or compromise subject safety.
* Subject has clinical evidence of recent major depression (by medical history) except those subjects already controlled by anti-depressants at screening.
* Subjects who, in the clinical judgement of the investigator, may be malingering or be motivated by secondary gain from participation in the study, will be excluded. Examples for consideration of exclusion include subjects who have compensation or social security claims pending in relation to their peripheral nerve injury or who are appealing against refusal of such claims, but subjects whose claims have been settled need not be excluded.
* Changes to medications permitted for the treatment of neuropathic pain within 4 weeks of the baseline period (Day -7), including dose adjustment, withdrawal of medications or initiation of new medications.
* Subjects who are unable to maintain the same medications for the treatment of neuropathic pain at the same stable dose as at baseline during the study.
* Unable to refrain from excessive use of sedative medications (e.g. benzodiazepines prescribed as hypnotics) that in the opinion of the Investigator may interfere with efficacy or safety assessments.
* Use of other prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication or during the study, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety or introduce a risk of drug-drug interactions.
* Unable to stop and remain abstain from non-pharmacological treatments for their neuropathic pain during the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the baseline period (Day -7) in the current study: 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of hypersensitivity to GW856553 or its components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within a 56 day period.
* Pregnant females as determined by positive urine or serum human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the study procedures
* Subject is mentally or legally incapacitated.
* Subjects with conditions requiring immunosuppressive therapy, or otherwise considered immunosuppressed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in average daily pain score from baseline to Week 4 of treatment based on the 11 point Pain Intensity Numerical Rating Scale (PI-NRS) | Baseline (Day -7) and Week 4
  The PI-NRS is an eleven point scale with 0=no pain and 10=worst pain imaginable. Participants rated the pain intensity for the neuropathic pain associated with the nerve injury and not pain from other concomitant causes. Change from baseline was calculated as endpoint value minus the baseline value.

SECONDARY OUTCOMES:
Change in average daily pain score from baseline to Weeks 1, 2 and 3 of treatment and the week before the follow-up visit | Baseline (Day -7) and up to Week 3
  The PI-NRS is an eleven point scale with 0=no pain and 10=worst pain imaginable. Participants rated the pain intensity for the neuropathic pain associated with the nerve injury and not pain from other concomitant causes. Change from baseline was calculated as endpoint value minus the baseline value.
Change from baseline in intensity of Dynamic Allodynia at Days 14 and 28 of treatment | Baseline (Day -7) and Day 14, 28
  Dynamic allodynia is a ten point scale with 0=no pain and 10=maximum pain. Intensity of dynamic allodynia was evaluated at the location of the participant's area of greatest tenderness related to the peripheral nerve injury. Change from baseline was calculated as endpoint value minus the baseline value.
Change from baseline in intensity of static hyperalgesia at Days 14 and 28 of treatment | Baseline (Day -7) and Day 14, 28
  The static hyperalgesia is an 10 point scale with 0=no pain and 10=maximum pain. Intensity of static mechanical hyperalgesia was evaluated at the location of the participant's area of greatest tenderness related to the peripheral nerve injury. Change from baseline was calculated as endpoint value minus the baseline value.
Change from baseline in pain quality on the Short-Form McGill Pain Questionnaire (SF-MPQ) at Days 14 and 28 of treatment and the follow-up visit | Baseline (Day -7) and Day 14, 28
  Each of 11 sensory and 4 affective descriptors were rated by the participant on a 4-point intensity scale (0 = none, 1 = mild, 2 = moderate and 3 = severe) and intensities were summed to provide sensory and affective scores, respectively. All 15 descriptors were used to calculate a total score. Change from baseline was calculated as endpoint value minus the baseline value.
Change from baseline in Galer Neuropathic Pain Scale to Days 14 and 28 of treatment and the follow-up visit | Baseline (Day -7), Day 14, 28 and follow-up (within approximately 14 days post Week 4)
  Each of 10 descriptors (2 that assess global dimensions of pain intensity and unpleasantness and 8 that assess specific qualities of neuropathic pain) were rated by the participant on an 11-point scale (0 = "no pain" or "not painful" and 10 = "the most painful sensation imaginable"). The ratings were added to provide a total score. Intent-to-Treat. Here, n= number of participants analyzed at particular time point.
Number of participants who have greater than or equal to (>=) 30 percent (%) and >=50% reduction in average daily pain score | Week 1, 2, 3, 4 and a week before follow-up (within approximately 14 days post Week 4)
  Data for participants who had >= 30 % and >=50% reduction in average daily pain score have been reported. Data for number of participants has been reported.
Number of Participants who have improved, much improved or very much improved relative to baseline on the Patient Global Impression of Change (PGIC) | Week 2, 4 and follow-up (within approximately 14 days post Week 4)
  PGIC assessed the change in overall status as perceived participant, respectively, according to a 7-point numerical rating scale (1- no change, 5-minimally worse, 6-much worse and 7, very much worse). Data for number of participants has been reported.very much improved, 2- much improved, 3-minimally improved, 4-
Number of Participants who have who have improved, much improved or very much improved relative to baseline on the Clinical Global Impression of Change (CGIC) | Week 2, Week 4 and follow-up(within approximately 14 days post Week 4)
  CGIC assessed the change in overall status as perceived by the clinician, according to a 7-point numerical rating scale (1- Very much improved, 2- much improved, 3- minimally improved, 4- no change, 5- minimally worse, 6- much worse and 7-very much worse).
Change from baseline in the amount of rescue medication used at Week 4 of treatment | Baseline (Day -7) and Week 4
  Any participant for whom the pain intensity became unacceptable during any stage of the study, including during washout period of prohibited analgesic medications, were permitted to initiate rescue analgesic therapy with paracetamol/acetaminophen up to a maximum dose of two 500 mg tablets two times daily (i.e., 2,000 mg per 24 hour period). Change from baseline is calculated as baseline value minus the endpoint value.
Change from baseline in total Profile of Mood States (POMS) score and POMS domains scores up to Week 2 and 4 of treatment | Baseline (Day -7), Week 2 and 4
  POMS is a list of 65 descriptors of mood that are each rated on a five point scale by subjects (0=applies not at all, 4=applies extremely) and that yield six scores: tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue inertia and confusion-bewilderment, as well as an overall mood disturbance score. Change from baseline is calculated as baseline value minus the endpoint value.
Change from baseline in SF-36 Health to Day 28 of treatment. | Baseline (Day -7) and Week 4
  The SF-36 is a subject-completed 36-item questionnaire used to evaluate participant's perception of their general quality of life in 8 areas: physical functioning, role physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role emotional (role limitations caused by emotional problems), vitality and general perception of health. Change from baseline is calculated as baseline value minus the endpoint value.
Number of participants with Adverse events (AEs) and Serious adverse events (SAEs) | Up to follow-up (within approximately 14 days post Week 4)
  An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Pre-dose and post-dose plasma GW856553 concentrations on Days 14 and 28 | Pre-dose (0 hour), 0-1, 1-2.5, 8-10, 10-12, 12-14 and 14-18 hours post-dose on Day 14 and 28
  Blood samples were withdrawn to analyze Pre-dose and post-dose plasma GW856553 concentrations on Pre-dose (0 hour), 0-1, 1-2.5, 8-10, 10-12, 12-14 and 14-18 hours post-dose on Day 14 and 28.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- Australia (2):
  - GSK Investigational Site, Broadmeadow, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
- Denmark (3):
  - GSK Investigational Site, Aarhus C
  - GSK Investigational Site, Koebenhavn NV
  - GSK Investigational Site, Odense C
- Norway (3):
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Trondheim
  - GSK Investigational Site, Tønsberg
- Russia (4):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Yaroslavl
- Spain (5):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Ourense
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Stockholm
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Thor Ostenfeld, Nathalie E. Richard, Alok Krishen, Robert Y. Lai, Jonathan Bullman, Amanda J. Baines, Joanne Green, Praveen Anand, Madeline Kelly . A randomised, double blind, placebo controlled study to evaluate the analgesic efficacy and safety of the novel p38 MAP kinase inhibitor, losmapimod, in patients with neuropathic pain following peripheral nerve injury . Eur J Pain. 2012;(Dec 14):
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register